CLINICAL TRIAL: NCT07278882
Title: A Randomized Controlled Trial of Mobile Technology-assisted Outpatient Maintenance Therapy in Children With Acute Lymphoblastic Leukaemia (ALL)
Brief Title: Using Mobile Technology-assisted Outpatient Maintenance Therapy Pediatric ALL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IIT2024105
Record Dates: First submitted 2025-11-18; First posted 2025-12-12 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12

CONDITIONS: Pediatric Acute Leukemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): A mobile application classifies each subject's maintenance therapy dosing status as 'On Track', 'Orange Alert', or 'Red Alert' based on analysis of his/her electronic diary of medication and blood tests.
  Interventions: Behavioral: Health monitoring & reminders for a mobile-phone portal for scheduling a telemedicine clinic visit and receive periodic model-phone messages instructing follow-up blood testing and dose adjustment.
- Control group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Health monitoring & reminders for a mobile-phone portal for scheduling a telemedicine clinic visit and receive periodic model-phone messages instructing follow-up blood testing and dose adjustment. — Subjects classified as 'Orange Alert' receive mobile-phone alert messages that instruct them to self-adjust dose of oral medication. Subjects classified as 'Red Alert' are directed to a mobile-phone portal for scheduling a telemedicine clinic visit and receive periodic model-phone messages instructing follow-up blood testing and dose adjustment.
  Arms: Intervention group

SUMMARY:
To assess the efficacy of using mobile technology to improve the percentage of time wherein drug dosing is within the target range

ELIGIBILITY:
Inclusion Criteria:

* 1) < 16 years old at diagnosis;
* 2) having demonstrated ≥ 3 months of > 90% compliance with using a mobile app to log in records of daily medication and weekly blood test results;
* 3) patient or legal guardian provides informed consent

Exclusion Criteria:

* None

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-11-20 (Estimated); Study Completion 2027-11-20 (Estimated)

PRIMARY OUTCOMES:
Percentage of time wherein white blood cell concentration is within the target range | After randomization
  Percentage of time wherein white blood cell concentration is within the target range 2.0 - 3.0 × 10^9/L after randomization.

SECONDARY OUTCOMES:
Percentage of time wherein white blood cell concentration is < 1.0 or > 5.0 × 10^9/L | After randomization
  Percentage of time wherein white blood cell concentration is < 1.0 or > 5.0 × 10^9/L after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

DOCUMENTS (1):
  • Study Protocol (2026-01-29): https://cdn.clinicaltrials.gov/large-docs/82/NCT07278882/Prot_001.pdf